CLINICAL TRIAL: NCT03207581
Title: RCT: Effect of Coaching on Mid-Career Physician Well-Being, Job Satisfaction, and Fulfillment
Brief Title: Effect of Coaching on Mid-Career Physician Well-Being, Job Satisfaction, and Fulfillment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Liselotte (Lotte) N. Dyrbye, Professor of Medicine and Medical Education, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17-003910
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Coaching Intervention (Experimental): Immediate Coaching Intervention arm will receive professional coaching
  Interventions: Behavioral: Professional Coaching
- Control/Delayed Coaching Intervention (Active Comparator): Participants randomized to the Control/Delayed Coaching will receive no intervention for the first six months of the study, at which point they cross over and receive 6 professional coaching sessions
  Interventions: Behavioral: Professional Coaching

INTERVENTIONS:
Behavioral: Professional Coaching — Professional, individualized coaching

SUMMARY:
The study will assess the effect of individualized professional coaching for mid-career family medicine and general internal medicine physicians on burnout, job satisfaction, and professional fulfillment.

ELIGIBILITY:
Inclusion Criteria

1. General internal medicine and family physicians
2. In practice for 5-30 years

Exclusion Criteria:

1. physicians who specialize in areas other than general internal medicine and family medicine
2. physicians who have been in practice less than 5 years or more than 30 years

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory score | 6 month
Change in Physician Job Satisfaction Scale score | 6 month
change in Empowerment at Work Scale score | 6 month
change in Utrecht Work Engagement score | 6 months

SECONDARY OUTCOMES:
Change in Maslach Burnout Inventory score | 12 month
Change in Physician Job Satisfaction Scale score | 12 months
change in Empowerment at Work Scale score | 12 months
change in Utrecht Work Engagement score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte N Dyrbye, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Dyrbye LN, Shanafelt TD, Gill PR, Satele DV, West CP. Effect of a Professional Coaching Intervention on the Well-being and Distress of Physicians: A Pilot Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1406-1414. doi: 10.1001/jamainternmed.2019.2425. PMID 31380892